CLINICAL TRIAL: NCT05481814
Title: The Role of Cardiopulmonary Stress Testing in Diagnostic Evaluation of Paradoxical Low Gradient Aortic Valve Stenosis
Brief Title: CPX in Paradoxical Low Flow Aortic Stenosis
Status: Withdrawn | Type: Observational
Why Stopped: Inability to execute internal logistics to begin enrollment
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Karthikeyan Ananthasubramaniam, Senior Staff Cardiologist, Henry Ford Health System
Other Study IDs: PLFLGAS1
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe aortic stenosis is a condition with poor life expectancy once it becomes symptomatic. There are no prospective studies illustrating the utility of cardiopulmonary stress (CPX) testing in diagnosing and prognosticating patients with paradoxically low gradient and low flow severe aortic stenosis. We aim to prospectively investigate the utility of CPX in this patient population with the hypothesis that utilizing CPX parameters would better identify higher risk patients warranting further evaluation and possibly intervention sooner.

DETAILED DESCRIPTION:
This will be a prospective crossectional, longitudinal study recruiting patients by invitation with paradoxical low flow low gradient severe aortic stenosis. Patients with PLFLG AS will have been identified in other studies and these patients will be approached for enrollment in the study. Patients deemed appropriate for enrollment will undergo recumbent bicycle stress testing with concomitant measure of gas exchange. The bicycle will be at 30 degrees with initiation of minimal resistance for 3 minutes, followed by an increase in work-rate of 25 watts every two minutes until the patient reaches a sign/symptom-limited maximum exertion or test limiting symptoms develop. Charts will be reviewed for baseline medical conditions and demographics. CPX protocol will be standard HFH protocol supervised by exercise physiologist. The first phase of the study will be investigating if these asymptomatic patients will be reclassified to symptomatic as defined by reduced V02 Max. The second phase will be following these patients for long term adverse events and if V02 max correlates with a higher risk.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve area <1 cm2
* Mean aortic pressure gradient <40 mmHg,
* Left ventricular ejection fraction >50% by 2D transthoracic echocardiography

Exclusion Criteria:

* Ischemic heart disease
* Severe mitral valve disease (regurgitation or stenosis)
* Moderate or severe aortic regurgitation
* Pulmonary hypertension (PA pressure >50 mmHg)
* COPD
* Uncontrolled hypertension (Systolic BP or Diastolic BP greater than 150/90)
* Inability or unwillingness to exercise.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with paradoxical low flow low gradient aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Functional status | August 30 2017-April 30 2017
  Evaluate changes in rest vs. Peak V02 at maximal exercise capacity.

SECONDARY OUTCOMES:
Follow-up | August 30 2017- August 30 2019
  Follow patients long term for major adverse cardiac events including myocardial infarction, stroke, hospitalization, or death and if CPX parameters provide further prognostic information in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Ananthasubramaniam, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States